CLINICAL TRIAL: NCT05248152
Title: Psychosocial and Psychophysical Factors Influencing the Effect of Preemptive Systemic Analgesia in Combination With Regional Anesthesia on Postoperative Pain Following Upper Limb Surgery
Brief Title: Effect of Psychosocial and Psychophysical Factors and Preemptive Analgesia on Postoperative Pain in Upper Limb Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Benjamin Jonke, Doctor of Medicine, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0120-182/2021/8
Record Dates: First submitted 2022-02-09; First posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen; Ibuprofen; Pregabalin

STUDY DESIGN:
Intervention Model Description: Three groups of patients with three different treatment regimens
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will receive either the actual drug or placebo. A separate investigator will be in charge of preparing the capsules and intravenous solutions that patients will receive before surgery in a way that it will not be possible to determine whether it is an actual drug or a placebo. That investigator will also write in which group the patient is on a piece of paper and insert it in the patient's inventory for safety purposes. The person that will measure the conditioned pain modulation and complete the pain questionnaires with patients will be a separate investigator. The anesthesiologist performing the axillary block will also be blinded, because the drugs/placebo will be prepared by a separate investigator. We will code the group to which the patients are allocated, so that the Outcomes Assessor will also be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Patients will receive a placebo capsule in the hour before surgery and two intravenous doses of saline before surgical incision.
  Interventions: Drug: Placebo
- Pregabalin (Experimental): Patients will receive pregabalin 150 mg in the hour before surgery and two intravenous doses of saline before surgical incision.
  Interventions: Drug: Pregabalin 150mg
- Paracetamol and Ibuprofen (Experimental): Patients will receive a placebo capsule in the hour before surgery and an intravenous dose of paracetamol 1 g and ibuprofen 400 mg before surgical incision.
  Interventions: Combination Product: Paracetamol and Ibuprofen

INTERVENTIONS:
Combination Product: Paracetamol and Ibuprofen — Patients will receive paracetamol 1g and ibuprofen 400 mg before surgical incision.
  Arms: Paracetamol and Ibuprofen
Drug: Pregabalin 150mg — Patients will receive pregabalin 150 mg in the hour before surgery
  Arms: Pregabalin
Drug: Placebo — Patients will receive a placebo capsule in the hour before surgery and two intravenous doses of saline before surgical incision.
  Arms: Placebo

SUMMARY:
The purpose of this study is to define the role of preemptive systemic analgesia in combination with regional anesthetic techniques on postoperative pain following upper limb surgery in different subgroups of patients with different psychosocial and psychophysical characteristics.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, patients will be given written informed consent. The study will include patients between the ages of 18 and 65, rated 1 or 2 by the American Society of Anesthesiologists (ASA) classification scheduled for distal radius surgery.

We will exclude patients with a known allergy to or adverse reaction to a local anesthetic, opioid, paracetamol or non-steroidal anti-inflammatory drugs, patients with a known opioid dependence, injection site infection, chronic pain, renal disease, known neuropathy, liver disease, with psychiatric disorders and diabetics.

The study will be randomized, prospective and double-blind. We will study the effect of preemptive dose of paracetamol and ibuprofen and pregabalin on postoperative pain after distal radius surgery in patients with different psychosocial and psychophysical characteristics. Patients will be admitted to the ward the day before surgery. At that time, we will explain to them the course of the research and offer them participation. For those with a written consent we will perform preoperative quantitative sensory tests on the same day and give them pain questionnaires.

We will determine conditional pain modulation by first applying a mechanical test stimulus of increasing intensity with an algometer to the skin of the volar side of the forearm and the skin in the middle of the front of the thigh contralateral to the injury until the patient experiences pain on the visual analog scale (VAS) 4/10. At that point the patients will press the patient operated button on the algometer and the stimulus will be stopped with the measurement stored. We will then repeat the same test together with a conditional stimulus - immersion of the ipsilateral lower extremity in cold water at 2 degrees Celsius. Conditional pain modulation will be calculated by subtracting the intensity of the independent primary stimulus from the intensity of the primary stimulus together with a concomitant conditioned stimulus. The end result will be the average of the values obtained on the skin of the volar side of the forearm and the skin in the middle of the front of the thigh.

On the same day the patients will also complete a Pain Catastrophising Scale (PCS) Questionnaire and a Brief Pain Inventory (BPI). They will also receive a short questionnaire to assess the pain and quality of sleep on the first night after surgery, which they will complete together with an anesthesiologist the morning after surgery.

On the day of surgery, patients will be divided into 3 groups:

The first group will receive pregabalin 150 mg per os 1 hour before arrival in the operating room and two intravenous doses of 100 ml of saline within 30 minutes before the surgical incision.

The second group will receive a placebo capsule per os 1 hour before arrival in the operating room and a preemptive intravenous dose of paracetamol 1 g and ibuprofen 400 mg within 30 minutes before the surgical incision.

The third group will receive a placebo capsule per os 1 hour before arrival in the operating room and two intravenous doses of 100 ml of saline within 30 minutes before the surgical incision.

All three groups will then receive an axillary block under ultrasound control by an experienced anesthesiologist. They may receive midazolam and/or fentanyl/sufentanil for anxiolysis and analgesia during the blockade. The surgery will be performed with of without sedation with propofol, titrated to desired effect. In the event of a failed block, patients will be placed under general anesthesia and excluded from the study. For postoperative nausea and vomiting they will not receive dexamethasone.

Postoperative analgesia:

For the postoperative analgesia, patients will receive a PCA (patient controlled analgesia) pump with Piritramide 45 mg diluted to 90 ml of saline. The PCA pump will have no continuous flow. The PCA boluses will be 3 mg every 20 minutes, with a 2 hour limit of 9 mg and a 6 hour limit of 15 mg. The PCA pump will be connected to the patients for at least 24 hours.

If necessary, the ward nurse will administer an additional intravenous dose of Piritramide 3 mg every 4 hours in case of insufficient analgesia (pain on VAS > 3/10). Patients will additionally receive intravenous Paracetamol 1 g every 6 h and intravenous Ibuprofen 400 mg every 8 hours.

For 24 hours after surgery we will record pain experienced by the patients, based on the VAS. Opioid consumption will be recorded by the PCA pump, any additional boluses by the nurses will be added to the total consumption. The first day after surgery, 14 days after surgery and 3 months after surgery the patients will again complete a BPI questionnaire. We will also document the interval between the injury and surgery, time of surgery, AO Distal Radius Fracture Classification, surgical approach and type of osteosynthesis.

We will study the impact of psychosocial, psychophysical and preemptive systemic analgesia on acute and chronic postoperative pain in distal radius surgery. We will examine whether patients with different psychosocial and psychophysical characteristics benefit differently from different regimens of preemptive systemic analgesia.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification score 1 and 2
* Patients with a distal radius fracture, scheduled for surgery

Exclusion Criteria:

* Allergy to a local anesthetic, opioid, paracetamol or a non-steroidal antirheumatic drug
* Opioid addiction
* Infection at the injection site
* Chronic pain syndromes
* Neuropathies
* Liver cirrhosis
* Chronic kidney disease stage 3 or higher
* Diabetes
* Psychiatric illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-01-13 (Actual); Primary Completion 2024-01-13 (Estimated); Study Completion 2024-04-13 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption in the first 24 hours | First 24 hours, starting at time of surgery
  Piritramide consumption will be obtained from the PCA pumb, manual boluses will be added.
Worst pain in the first 24 hours | First 24 hours, starting at time of surgery
  Worst pain in the first 24 hours after surgery on the visual analog scale (VAS) will be obtained the day after surgery

SECONDARY OUTCOMES:
The incidence of chronic pain | Three months after surgery
  The presence of chronic pain will be defined as pain persisting at the three month interval
Sleep quality on the night after surgery | First 24 hours, starting at time of surgery
  Sleep quality will be obtained by a questionnaire, raging from 1-5, where 1 is described as very poor sleep quality and 5 as very good sleep quality
Opioid consumption in the first 24 hours in correlation with preoperative Pain catastrophising scale (PCS) | First 24 hours, starting at time of surgery
  PCS will be obtained preoperatively, we will investigate, whether there is a positive correlation between opioid consumption in the first 24 hours and preoperative PCS greater than 30. PCS is a questionnaire, consisting of 13 questions, each ranging from scores 0 to 4, so the final score is in the range of 0 to 52. A total PCS score of 30 or more represents clinically relevant level of pain catastrophizing.
Worst pain in the first 24 hours in correlation with preoperative Pain catastrophising scale (PCS) | First 24 hours, starting at time of surgery
  PCS will be obtained preoperatively, we will investigate, whether there is a positive correlation between the worst pain in the first 24 hours and preoperative PCS greater than 30. PCS is a questionnaire, consisting of 13 questions, each ranging from scores 0 to 4, so the final score is in the range of 0 to 52. A total PCS score of 30 or more represents clinically relevant level of pain catastrophizing.
Opioid consumption in the first 24 hours in correlation with preoperative Conditioned pain modulation (CPM) | First 24 hours, starting at time of surgery
  CPM will be obtained preoperatively, we will investigate, whether there is a correlation between opioid consumption in the first 24 hours and preoperative CPM. CPM will be determined by first applying a mechanical test stimulus of increasing intensity with an algometer to the skin of the volar side of the forearm and the skin in the middle of the front of the thigh contralateral to the injury until the patient experiences pain on the visual analog scale (VAS) of 4/10. The same stimulus will then be applied together with a conditional stimulus - immersion of the ipsilateral lower extremity in cold water at 2 degrees Celsius. Conditional pain modulation will be calculated by subtracting the intensity of the independent primary stimulus from the intensity of the primary stimulus together with a concomitant conditioned stimulus. CPM is a centrally processed measure of the net effect of the descending pain pathway. Higher CPM scores signify better pain control.
Worst pain in the first 24 hours in correlation with preoperative Conditioned pain modulation (CPM) | First 24 hours, starting at time of surgery
  CPM will be obtained preoperatively, we will investigate, whether there is a correlation between the worst pain in the first 24 hours and preoperative CPM. CPM will be determined by first applying a mechanical test stimulus of increasing intensity with an algometer to the skin of the volar side of the forearm and the skin in the middle of the front of the thigh contralateral to the injury until the patient experiences pain on the visual analog scale (VAS) of 4/10. The same stimulus will then be applied together with a conditional stimulus - immersion of the ipsilateral lower extremity in cold water at 2 degrees Celsius. Conditional pain modulation will be calculated by subtracting the intensity of the independent primary stimulus from the intensity of the primary stimulus together with a concomitant conditioned stimulus. CPM is a centrally processed measure of the net effect of the descending pain pathway. Higher CPM scores signify better pain control.
The incidence of chronic pain in correlation with preoperative Conditioned pain modulation (CPM) | 3 months after surgery
  CPM will be obtained preoperatively, we will investigate, whether there is a correlation between the incidence of chronic pain at three months after surgery and preoperative CPM. CPM will be determined by first applying a mechanical test stimulus of increasing intensity with an algometer to the skin of the volar side of the forearm and the skin in the middle of the front of the thigh contralateral to the injury until the patient experiences pain on the visual analog scale (VAS) of 4/10. The same stimulus will then be applied together with a conditional stimulus - immersion of the ipsilateral lower extremity in cold water at 2 degrees Celsius. Conditional pain modulation will be calculated by subtracting the intensity of the independent primary stimulus from the intensity of the primary stimulus together with a concomitant conditioned stimulus. CPM is a centrally processed measure of the net effect of the descending pain pathway. Higher CPM scores signify better pain control.
The incidence of chronic pain in correlation with preoperative Pain catastrophising scale (PCS) | 3 months after surgery
  PCS will be obtained preoperatively, we will investigate, whether there is a positive correlation between the incidence of chronic pain at three months after surgery and preoperative PCS greater than 30. PCS is a questionnaire, consisting of 13 questions, each ranging from scores 0 to 4, so the final score is in the range of 0 to 52. A total PCS score of 30 or more represents clinically relevant level of pain catastrophizing.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Jonke, M.D., Principal Investigator — University Medical Centre Ljubljana
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
We will include all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the data.

REFERENCES:
- [Background] Hewson DW, Oldman M, Bedforth NM. Regional anaesthesia for shoulder surgery. BJA Educ. 2019 Apr;19(4):98-104. doi: 10.1016/j.bjae.2018.12.004. Epub 2019 Feb 6. No abstract available. PMID 33456877
- [Background] Hadzic A, Williams BA, Karaca PE, Hobeika P, Unis G, Dermksian J, Yufa M, Thys DM, Santos AC. For outpatient rotator cuff surgery, nerve block anesthesia provides superior same-day recovery over general anesthesia. Anesthesiology. 2005 May;102(5):1001-7. doi: 10.1097/00000542-200505000-00020. PMID 15851888
- [Background] Dunkman WJ, Manning MW. Enhanced Recovery After Surgery and Multimodal Strategies for Analgesia. Surg Clin North Am. 2018 Dec;98(6):1171-1184. doi: 10.1016/j.suc.2018.07.005. Epub 2018 Aug 22. PMID 30390850
- [Background] Nimmo SM, Foo ITH, Paterson HM. Enhanced recovery after surgery: Pain management. J Surg Oncol. 2017 Oct;116(5):583-591. doi: 10.1002/jso.24814. Epub 2017 Sep 5. PMID 28873505
- [Background] Simpson JC, Bao X, Agarwala A. Pain Management in Enhanced Recovery after Surgery (ERAS) Protocols. Clin Colon Rectal Surg. 2019 Mar;32(2):121-128. doi: 10.1055/s-0038-1676477. Epub 2019 Feb 28. PMID 30833861
- [Background] Wick EC, Grant MC, Wu CL. Postoperative Multimodal Analgesia Pain Management With Nonopioid Analgesics and Techniques: A Review. JAMA Surg. 2017 Jul 1;152(7):691-697. doi: 10.1001/jamasurg.2017.0898. PMID 28564673
- [Background] Rosero EB, Joshi GP. Preemptive, preventive, multimodal analgesia: what do they really mean? Plast Reconstr Surg. 2014 Oct;134(4 Suppl 2):85S-93S. doi: 10.1097/PRS.0000000000000671. PMID 25255012
- [Background] Kelly DJ, Ahmad M, Brull SJ. Preemptive analgesia I: physiological pathways and pharmacological modalities. Can J Anaesth. 2001 Nov;48(10):1000-10. doi: 10.1007/BF03016591. PMID 11698320
- [Background] Doleman B, Read D, Lund JN, Williams JP. Preventive Acetaminophen Reduces Postoperative Opioid Consumption, Vomiting, and Pain Scores After Surgery: Systematic Review and Meta-Analysis. Reg Anesth Pain Med. 2015 Nov-Dec;40(6):706-12. doi: 10.1097/AAP.0000000000000311. PMID 26469366
- [Background] Ong CK, Lirk P, Seymour RA, Jenkins BJ. The efficacy of preemptive analgesia for acute postoperative pain management: a meta-analysis. Anesth Analg. 2005 Mar;100(3):757-773. doi: 10.1213/01.ANE.0000144428.98767.0E. PMID 15728066
- [Background] Wang K, Luo J, Zheng L, Luo T. Preoperative flurbiprofen axetil administration for acute postoperative pain: a meta-analysis of randomized controlled trials. J Anesth. 2017 Dec;31(6):852-860. doi: 10.1007/s00540-017-2409-0. Epub 2017 Sep 21. PMID 28936554
- [Background] Esparza-Villalpando V, Pozos-Guillen A, Masuoka-Ito D, Gaitan-Fonseca C, Chavarria-Bolanos D. Analgesic efficacy of preoperative dexketoprofen trometamol: A systematic review and meta-analysis. Drug Dev Res. 2018 Mar;79(2):47-57. doi: 10.1002/ddr.21419. Epub 2017 Dec 15. PMID 29243848
- [Background] Ong CK, Seymour RA, Lirk P, Merry AF. Combining paracetamol (acetaminophen) with nonsteroidal antiinflammatory drugs: a qualitative systematic review of analgesic efficacy for acute postoperative pain. Anesth Analg. 2010 Apr 1;110(4):1170-9. doi: 10.1213/ANE.0b013e3181cf9281. Epub 2010 Feb 8. PMID 20142348
- [Background] Mishriky BM, Waldron NH, Habib AS. Impact of pregabalin on acute and persistent postoperative pain: a systematic review and meta-analysis. Br J Anaesth. 2015 Jan;114(1):10-31. doi: 10.1093/bja/aeu293. Epub 2014 Sep 10. PMID 25209095
- [Background] Calandre EP, Rico-Villademoros F, Slim M. Alpha2delta ligands, gabapentin, pregabalin and mirogabalin: a review of their clinical pharmacology and therapeutic use. Expert Rev Neurother. 2016 Nov;16(11):1263-1277. doi: 10.1080/14737175.2016.1202764. Epub 2016 Jul 7. PMID 27345098
- [Background] Khalili G, Janghorbani M, Saryazdi H, Emaminejad A. Effect of preemptive and preventive acetaminophen on postoperative pain score: a randomized, double-blind trial of patients undergoing lower extremity surgery. J Clin Anesth. 2013 May;25(3):188-92. doi: 10.1016/j.jclinane.2012.09.004. Epub 2013 Apr 6. PMID 23567482
- [Background] Boonriong T, Tangtrakulwanich B, Glabglay P, Nimmaanrat S. Comparing etoricoxib and celecoxib for preemptive analgesia for acute postoperative pain in patients undergoing arthroscopic anterior cruciate ligament reconstruction: a randomized controlled trial. BMC Musculoskelet Disord. 2010 Oct 25;11:246. doi: 10.1186/1471-2474-11-246. PMID 20973952
- [Background] Wang J, Li H, Ma H, Wang N. Effect of Preemptive Flurbiprofen Axetil and Tramadol on Transurethral Resection of the Prostate under Spinal Anesthesia. Pain Res Treat. 2016;2016:3942040. doi: 10.1155/2016/3942040. Epub 2016 Feb 9. PMID 26977315
- [Background] Khezri MB, Mosallaei MA, Ebtehaj M, Mohammadi N. Comparison of preemptive effect of intravenous ketorolac versus meperidine on postoperative shivering and pain in patients undergoing cesarean section under spinal anesthesia: A prospective, randomized, double-blind study. Caspian J Intern Med. 2018 Spring;9(2):151-157. doi: 10.22088/cjim.9.2.151. PMID 29732033
- [Background] Demir U, Ince I, Aksoy M, Dostbil A, Ari MA, Sulak MM, Kose M, Tanios M, Ozmen O. The Effect of Pre-emptive Dexketoprofen Administration on Postoperative Pain Management in Patients with Ultrasound Guided Interscalene Block in Arthroscopic Shoulder Surgery. J Invest Surg. 2021 Jan;34(1):82-88. doi: 10.1080/08941939.2019.1576809. Epub 2019 Apr 9. PMID 30966835
- [Background] Park M, Lee H, Jeon Y. Preoperative pregabalin prolongs duration of spinal anesthesia and reduces early postoperative pain: A double-blind, randomized clinical CONSORT study. Medicine (Baltimore). 2016 Sep;95(36):e4828. doi: 10.1097/MD.0000000000004828. PMID 27603398
- [Background] Akhavanakbari G, Entezariasl M, Isazadehfar K, Mirzarahimi T. The effects of oral pregabalin on post-operative pain of lower limb orthopedic surgery: A double-blind, placebo-controlled trial. Perspect Clin Res. 2013 Jul;4(3):165-8. doi: 10.4103/2229-3485.115376. PMID 24010057
- [Background] Bafna U, Rajarajeshwaran K, Khandelwal M, Verma AP. A comparison of effect of preemptive use of oral gabapentin and pregabalin for acute post-operative pain after surgery under spinal anesthesia. J Anaesthesiol Clin Pharmacol. 2014 Jul;30(3):373-7. doi: 10.4103/0970-9185.137270. PMID 25190946
- [Background] Omara AF, Ahmed SA, Abusabaa MM. The Effect Of The Use Of Pre-Emptive Oral Pregabalin On The Postoperative Spinal Analgesia In Patients Presented For Orthopedic Surgeries: Randomized Controlled Trial. J Pain Res. 2019 Sep 30;12:2807-2814. doi: 10.2147/JPR.S216184. eCollection 2019. PMID 31686901
- [Background] Cegin MB, Soyoral L, Yuzkat N, Baydi V, Goktas U. Pregabalin administered as an anxiolytic agent in ultrasound-guided infraclavicular block: a controlled, double-blind, dose-ranging trial. Eur Rev Med Pharmacol Sci. 2016;20(3):568-74. PMID 26914135
- [Background] Gatchel RJ, McGeary DD, McGeary CA, Lippe B. Interdisciplinary chronic pain management: past, present, and future. Am Psychol. 2014 Feb-Mar;69(2):119-30. doi: 10.1037/a0035514. PMID 24547798
- [Background] Tuna T, Boz S, Van Obbergh L, Lubansu A, Engelman E. Comparison of the Pain Sensitivity Questionnaire and the Pain Catastrophizing Scale in Predicting Postoperative Pain and Pain Chronicization After Spine Surgery. Clin Spine Surg. 2018 Nov;31(9):E432-E440. doi: 10.1097/BSD.0000000000000694. PMID 30036209
- [Background] Wright D, Hoang M, Sofine A, Silva JP, Schwarzkopf R. Pain catastrophizing as a predictor for postoperative pain and opiate consumption in total joint arthroplasty patients. Arch Orthop Trauma Surg. 2017 Dec;137(12):1623-1629. doi: 10.1007/s00402-017-2812-x. Epub 2017 Oct 3. PMID 28975493
- [Background] Granot M, Ferber SG. The roles of pain catastrophizing and anxiety in the prediction of postoperative pain intensity: a prospective study. Clin J Pain. 2005 Sep-Oct;21(5):439-45. doi: 10.1097/01.ajp.0000135236.12705.2d. PMID 16093750
- [Background] Khan RS, Skapinakis P, Ahmed K, Stefanou DC, Ashrafian H, Darzi A, Athanasiou T. The association between preoperative pain catastrophizing and postoperative pain intensity in cardiac surgery patients. Pain Med. 2012 Jun;13(6):820-7. doi: 10.1111/j.1526-4637.2012.01386.x. Epub 2012 May 8. PMID 22568812
- [Background] Burns LC, Ritvo SE, Ferguson MK, Clarke H, Seltzer Z, Katz J. Pain catastrophizing as a risk factor for chronic pain after total knee arthroplasty: a systematic review. J Pain Res. 2015 Jan 5;8:21-32. doi: 10.2147/JPR.S64730. eCollection 2015. PMID 25609995
- [Background] Treede RD. The role of quantitative sensory testing in the prediction of chronic pain. Pain. 2019 May;160 Suppl 1:S66-S69. doi: 10.1097/j.pain.0000000000001544. PMID 31008852
- [Background] Schreiber KL, Zinboonyahgoon N, Xu X, Spivey T, King T, Dominici L, Partridge A, Golshan M, Strichartz G, Edwards RR. Preoperative Psychosocial and Psychophysical Phenotypes as Predictors of Acute Pain Outcomes After Breast Surgery. J Pain. 2019 May;20(5):540-556. doi: 10.1016/j.jpain.2018.11.004. Epub 2018 Nov 23. PMID 30476655
- [Background] van Helmond N, Aarts HM, Timmerman H, Olesen SS, Drewes AM, Wilder-Smith OH, Steegers MA, Vissers KC. Is Preoperative Quantitative Sensory Testing Related to Persistent Postsurgical Pain? A Systematic Literature Review. Anesth Analg. 2020 Oct;131(4):1146-1155. doi: 10.1213/ANE.0000000000004871. PMID 32925335
- [Background] Sangesland A, Storen C, Vaegter HB. Are preoperative experimental pain assessments correlated with clinical pain outcomes after surgery? A systematic review. Scand J Pain. 2017 Apr;15:44-52. doi: 10.1016/j.sjpain.2016.12.002. Epub 2016 Dec 19. PMID 28850344
- [Background] Fernandes C, Pidal-Miranda M, Samartin-Veiga N, Carrillo-de-la-Pena MT. Conditioned pain modulation as a biomarker of chronic pain: a systematic review of its concurrent validity. Pain. 2019 Dec;160(12):2679-2690. doi: 10.1097/j.pain.0000000000001664. PMID 31365469
- [Background] Arendt-Nielsen L, Egsgaard LL, Petersen KK, Eskehave TN, Graven-Nielsen T, Hoeck HC, Simonsen O. A mechanism-based pain sensitivity index to characterize knee osteoarthritis patients with different disease stages and pain levels. Eur J Pain. 2015 Nov;19(10):1406-17. doi: 10.1002/ejp.651. Epub 2014 Dec 29. PMID 25545011
- [Background] Petersen KK, Graven-Nielsen T, Simonsen O, Laursen MB, Arendt-Nielsen L. Preoperative pain mechanisms assessed by cuff algometry are associated with chronic postoperative pain relief after total knee replacement. Pain. 2016 Jul;157(7):1400-1406. doi: 10.1097/j.pain.0000000000000531. PMID 27331347